CLINICAL TRIAL: NCT00005295
Title: Idiopathic Pulmonary Fibrosis: a Case-control Study
Status: Terminated | Type: Observational
Why Stopped: Not a clinical Trial & inadvertently entered in the system.
Sponsor: University of New Mexico (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 2018; R01HL043153 (NIH)
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Lung Diseases; Pulmonary Fibrosis; Lung Diseases, Interstitial
MeSH Terms: conditions — Lung Diseases; Pulmonary Fibrosis; Lung Diseases, Interstitial

SUMMARY:
To determine risk factors for idiopathic pulmonary fibrosis.

DETAILED DESCRIPTION:
BACKGROUND:

Idiopathic pulmonary fibrosis is a progressive and generally fatal disease that causes fibrosis of the pulmonary interstitium. While many environmental agents cause diseases clinically similar, the etiology of idiopathic pulmonary fibrosis suggests that environmental agents could incite the tissue injury that results in the disease; furthermore, host characteristics could have an important role in determining the magnitude of the host response to the agent initiating injury.

DESIGN NARRATIVE:

In this case control study, cases were ascertained at the multiple collaborating centers and controls were identified by telephone screening. A telephone interview was conducted to collect information needed to test hypotheses concerning cigarette smoking, occupational exposure, indoor exposures, other environmental factors, and host factors. To limit disease misclassification, two pathologists experienced with interstitial diseases of the lung reviewed histopathological material from all cases to exclude entities other than interstitial lung fibrosis and to fully characterize the cases clinically. The mortality of this large series of cases was also described.

ELIGIBILITY:
No eligibility criteria

Ages: 0 Years to 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1989-07; Study Completion 1995-06

REFERENCES:
- [Background] Baumgartner KB, Samet JM, Stidley CA, Colby TV, Waldron JA. Cigarette smoking: a risk factor for idiopathic pulmonary fibrosis. Am J Respir Crit Care Med. 1997 Jan;155(1):242-8. doi: 10.1164/ajrccm.155.1.9001319.
- [Background] Coultas DB, Gong H Jr, Grad R, Handler A, McCurdy SA, Player R, Rhoades ER, Samet JM, Thomas A, Westley M. Respiratory diseases in minorities of the United States. Am J Respir Crit Care Med. 1994 Mar;149(3 Pt 2):S93-131. doi: 10.1164/ajrccm/149.3_Pt_2.S93. No abstract available. PMID 8118656